CLINICAL TRIAL: NCT04362124
Title: Performance Evaluation of BCG Vaccination in Healthcare Personnel to Reduce the Severity of SARS-COV-2 Infection in Medellín, Colombia, 2020
Brief Title: Performance Evaluation of BCG Vaccination in Healthcare Personnel to Reduce the Severity of COVID-19 Infection.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was stopped because Principal Investigator did not obtain sponsorship to carry it out
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PEC03_2020
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: coronavirus; BCG; COVID-19; SARS-COV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: A multicenter, double-blind, randomized, phase III clinical trial, divided into two groups (vaccine and placebo) using a 1: 1 allocation ratio.
  The treatment allocation will be performed according to random code.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind trial. The blinding of the investigational vaccine will be maintained using an opaque label for the two products (vaccine and placebo).
  The subjects, who collect the data (e.g., investigator and coordinator) and who evaluate the data (e.g., statistician) will be blinded. One or more pharmacists/vaccine administrators designated from the facility will not be blinded. These designated unblinded individuals will maintain the blindness of the investigational vaccine and will not be involved in evaluating the safety of the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vaccine BCG (Experimental): A single dose intradermal application of 0.1 ml of between 1 x 105 to 33 x 105 CFU of BCG, in the deltoid of the non-dominant arm.
  Follow-up of the participant up to day 360. The frequency and intensity of possible Adverse Events, reactions, and symptoms that appear, and other reactions stipulated in the protocol will be documented in the subject's diary.
  Interventions: Biological: vaccine BCG
- Placebo (Placebo Comparator): A single dose intradermal application of 0.1ml of normal saline solution, in the deltoid of the non-dominant arm.
  Follow-up of the participant up to day 360. The frequency and intensity of possible Adverse Events, reactions, and symptoms that appear, and other reactions stipulated in the protocol will be documented in the subject's diary.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: vaccine BCG — Performance evaluation of a single dose of BCG vaccine in reducing the severity of SARS-COV-2 infection compared to placebo, in healthcare personnel.
  Other Names: BCG Liofilizada
  Arms: vaccine BCG
Other: Placebo — A single dose intradermal application of normal saline solution.
  Arms: Placebo

SUMMARY:
Until the first half of April, Colombia has more than 2,800 infected cases and a hundred deaths as a result of COVID-19, with Antioquia being the third department with the highest number of cases. Official records indicate that, in Colombia, the first case was diagnosed on March 6, 2020, corresponding to a patient from Italy. However, in conversations with several infectologists and intensivists from Medellín, it was agreed that clinical cases similar to the clinical presentation that is now recognized as COVID-19 had arisen since the end of 2019 when it was still unknown to everyone. The previous suggests that the virus was already circulating in the country since before March 6, 2020. But at that moment, there were no tools to make a clinical identification, nor to diagnose it from the laboratory's point of view.

Considering as real the hypothesis that the infection has been circulating in the country since before the first official diagnosis, the question arises: Why does not the country still has the same healthcare and humanitarian chaos that countries such as Italy and Spain are suffering at this time? To answer this question may be that there are differences in vaccination rates with BCG (Bacille Calmette-Guérin or tuberculosis vaccine), which is significantly higher in Latin America compared to those in Europe. This finding could explain to some extent the situation in the country, since previous studies have shown the influence that this vaccine can have on the immune response against various other pathogens, including viruses.

Among the population at risk of infection, health-care workers due to their permanent contact with patients are the population group with the highest risk of contracting SARS-Cov-2 and developing COVID-19 in any of its clinical manifestations, and currently there are no vaccines or proven preventive interventions available to protect them.

For this reason, this research study aims to demonstrate whether the centennial vaccine against tuberculosis (BCG), a bacterial disease, can activate the human immune system in a broad way, allowing it to better combat the coronavirus that causes COVID-19 and, perhaps, prevents the complications that lead the patient to the intensive care unit and death.

In the future, and if these results are as expected, they may be the basis for undertaking a population vaccination campaign that improves clinical outcomes in the general population.

DETAILED DESCRIPTION:
Problem Statement

To date, Colombia has more than 2,800 infected cases and a hundred deaths as a result of COVID-19, with Antioquia being the third department with the highest number of cases (1). Official records indicate that, in Colombia, the first case was diagnosed on March 6, 2020, corresponding to a patient from Italy. However, in conversations with several infectologists and intensivists from Medellín, it was agreed that clinical cases similar to the clinical presentation that is now recognized as COVID-19 had arisen since the end of 2019 when it was still unknown to everyone. The previous suggests that the virus was already circulating in the country since before March 6, 2020. But at that moment, there were no tools to make a clinical identification, nor to diagnose it from the laboratory's point of view. This theory has been gathering momentum in other latitudes, demonstrating how the asymptomatic infected individuals are responsible for spreading the infection .

Considering as real the hypothesis that the infection has been circulating in the country since before the first official diagnosis, the question arises: Why does not the country still has the same healthcare and humanitarian chaos that countries such as Italy and Spain are suffering at this time? To answer this question, an extensive literature search of factors that differentiate Europeans from Latin Americans was carried out. Finding, in addition to genetic factors specific to race, differences in the number of ACEI receptors (binding site of the coronavirus to the alveolus), and differences in vaccination rates with BCG (Bacille Calmette-Guérin or tuberculosis vaccine), which is significantly higher in Latin America compared to those in Europe (3). This last finding could explain to some extent the situation in the country, since previous studies have shown the influence that this vaccine can have on the immune response against various other pathogens, including viruses (4,5).

Among the population at risk of infection, health-care workers due to their permanent contact with patients are the population group with the highest risk of contracting SARS-Cov-2 and developing COVID-19 in any of its clinical manifestations.

Currently, there are no vaccines or proven preventive interventions available to protect health-care workers. However, researchers from Germany, the Netherlands, Australia, and France are working on a clinical trial with an unorthodox approach to combat this new virus. This research study aims to demonstrate whether the centennial vaccine against tuberculosis (BCG), a bacterial disease, can activate the human immune system in a broad way, allowing it to better combat the coronavirus that causes COVID-19 and, perhaps, prevents the complications that lead the patient to the intensive care unit and death. Initially, studies in these four countries will be carried out on doctors and nurses, since they are the ones with a higher risk of becoming infected compared to the general population.

Currently, the available evidence supports the hypothesis that BCG vaccination has beneficial heterologous effects against viral, bacterial, and fungal infections. The basis of these effects has been little explored in humans; however, this knowledge opens the door to future research to explore the effect of "trained immunity" associated with this vaccine, both for diseases in hosts with immunological disorders, and for autoinflammatory diseases, in which there is an inappropriate activation of inflammation (21). All of the findings described have considerable potential to aid in the design of new therapeutic strategies, such as the use of old and new vaccines that combine classical immune memory, and the activation of innate immunity by "trained immunity," for prevention and treatment of infections, and modulation of exaggerated inflammation in autoinflammatory diseases.

A multicenter, double-blind, randomized, phase III clinical trial will be carried out. 1000 healthy healthcare workers (doctors, nurses, and nursing assistants) with a negative test for COVID-19 and asymptomatic for the disease will be randomly assigned to receive one dose of BGC vaccine or placebo (saline solution). Volunteers will be followed for one year.

Hypothesis Healthcare workers who have negative SARS-Cov-2 serology and who receive the BCG vaccine, have a better clinical outcome if they become infected with COVID-19, in terms of not getting sick, requiring hospitalization or dying, than those who do not receive the vaccine.

Objectives

Overall Objective

Evaluate the performance of BCG vaccination in reducing the severity of SARS-COV-2 infection compared to the placebo, in healthcare personnel from Medellín, Colombia.

. Specific Objectives

* Determine if there are differences in the clinical outcome in terms of not getting sick, requiring hospitalization, or dying in both treatment groups.
* Estimate previous exposure of healthcare personnel to SARS-Cov-2 by conducting rapid tests that measure IgG and IgM immunity.
* Assess the safety (frequency, seriousness, and severity of adverse events) of BCG vaccination in an adult population.
* Estimate SARS-Cov-2 infection in healthcare personnel at the end of the study, by performing rapid tests that measure IgG and IgM immunity.

ELIGIBILITY:
Inclusion criteria

* Men and women
* Between ≥18 and ≤ 65 years old
* Healthcare workers (doctors, nurses and nursing assistants) from clinics and hospitals in Medellín, who are directly involved in the care of patients with COVID-19
* A negative test for COVID-19 and being asymptomatic at baseline
* Are able and willing to give signed informed consent (Subjects whom the investigator believes are able to understand and are willing to comply with the requirements of the protocol)

Exclusion Criteria

* Have a previous diagnosis (probable or confirmed) of COVID-19
* Immunosuppression (pharmacological or clinical)
* Are taking immunosuppressive medications
* Pregnant or lactating women; or women of childbearing age who do not agree to take contraceptives during the month following vaccination.
* Have received any live or replicative vaccine one month before the time of screening.
* Permanent teleworking activity.
* History of active tuberculosis
* Currently are receiving Hydroxychloroquine, Chloroquine, Lopinavir/ritonavir, Tocilizumab, or Azithromycin.
* Known or suspected history of hypersensitivity to vaccines.
* Patients who do not wish to attend or who cannot keep up with the follow-up visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | From date of randomization to 360 day of the study
  Incidence of COVID-19 cases confirmed or probable in the study population

SECONDARY OUTCOMES:
Secondary outcome | From date to diagnosis to 1 month after
  Incidence of severe or critical infection in COVID-19 cases
Secondary outcome | From date to diagnosis to 1 month after
  Lethality of the infection in both groups
Secondary outcome | From date of randomization to 7 day of the study
  Assess the safety (frequency, seriousness, and severity of adverse events) of BCG vaccination
Secondary outcome | At baseline evaluation
  Prevalence of SARS-Cov-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: Juan C cataño, MD.MI.ID, Principal Investigator — infectious medicine doctor
Locations (1):
- Program for Research and Control in Tropical Diseases - PECET, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li R, Pei S, Chen B, Song Y, Zhang T, Yang W, Shaman J. Substantial undocumented infection facilitates the rapid dissemination of novel coronavirus (SARS-CoV-2). Science. 2020 May 1;368(6490):489-493. doi: 10.1126/science.abb3221. Epub 2020 Mar 16. PMID 32179701
- [Background] Zwerling A, Behr MA, Verma A, Brewer TF, Menzies D, Pai M. The BCG World Atlas: a database of global BCG vaccination policies and practices. PLoS Med. 2011 Mar;8(3):e1001012. doi: 10.1371/journal.pmed.1001012. Epub 2011 Mar 22. PMID 21445325
- [Background] Arts RJW, Moorlag SJCFM, Novakovic B, Li Y, Wang SY, Oosting M, Kumar V, Xavier RJ, Wijmenga C, Joosten LAB, Reusken CBEM, Benn CS, Aaby P, Koopmans MP, Stunnenberg HG, van Crevel R, Netea MG. BCG Vaccination Protects against Experimental Viral Infection in Humans through the Induction of Cytokines Associated with Trained Immunity. Cell Host Microbe. 2018 Jan 10;23(1):89-100.e5. doi: 10.1016/j.chom.2017.12.010. PMID 29324233
- [Background] Moorlag SJCFM, Arts RJW, van Crevel R, Netea MG. Non-specific effects of BCG vaccine on viral infections. Clin Microbiol Infect. 2019 Dec;25(12):1473-1478. doi: 10.1016/j.cmi.2019.04.020. Epub 2019 May 2. PMID 31055165
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Benn CS, Netea MG, Selin LK, Aaby P. A small jab - a big effect: nonspecific immunomodulation by vaccines. Trends Immunol. 2013 Sep;34(9):431-9. doi: 10.1016/j.it.2013.04.004. Epub 2013 May 14. PMID 23680130
- [Background] Jensen KJ, Larsen N, Biering-Sorensen S, Andersen A, Eriksen HB, Monteiro I, Hougaard D, Aaby P, Netea MG, Flanagan KL, Benn CS. Heterologous immunological effects of early BCG vaccination in low-birth-weight infants in Guinea-Bissau: a randomized-controlled trial. J Infect Dis. 2015 Mar 15;211(6):956-67. doi: 10.1093/infdis/jiu508. Epub 2014 Sep 9. PMID 25210141
- [Background] Kleinnijenhuis J, van Crevel R, Netea MG. Trained immunity: consequences for the heterologous effects of BCG vaccination. Trans R Soc Trop Med Hyg. 2015 Jan;109(1):29-35. doi: 10.1093/trstmh/tru168. PMID 25573107
- [Background] Uthayakumar D, Paris S, Chapat L, Freyburger L, Poulet H, De Luca K. Non-specific Effects of Vaccines Illustrated Through the BCG Example: From Observations to Demonstrations. Front Immunol. 2018 Dec 4;9:2869. doi: 10.3389/fimmu.2018.02869. eCollection 2018. PMID 30564249
- [Background] Tribouley J, Tribouley-Duret J, Appriou M. [Effect of Bacillus Callmette Guerin (BCG) on the receptivity of nude mice to Schistosoma mansoni]. C R Seances Soc Biol Fil. 1978;172(5):902-4. French. PMID 157204
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Benn CS, Joosten LA, Jacobs C, van Loenhout J, Xavier RJ, Aaby P, van der Meer JW, van Crevel R, Netea MG. Long-lasting effects of BCG vaccination on both heterologous Th1/Th17 responses and innate trained immunity. J Innate Immun. 2014;6(2):152-8. doi: 10.1159/000355628. Epub 2013 Oct 30. PMID 24192057
- [Background] Sher NA, Chaparas SD, Greenberg LE, Bernard S. Effects of BCG, Corynebacterium parvum, and methanol-extration residue in the reduction of mortality from Staphylococcus aureus and Candida albicans infections in immunosuppressed mice. Infect Immun. 1975 Dec;12(6):1325-30. doi: 10.1128/iai.12.6.1325-1330.1975. PMID 1107224
- [Background] Sakuma T, Suenaga T, Yoshida I, Azuma M. Mechanisms of enhanced resistance of Mycobacterium bovis BCG-treated mice to ectromelia virus infection. Infect Immun. 1983 Nov;42(2):567-73. doi: 10.1128/iai.42.2.567-573.1983. PMID 6315580
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Joosten LA, Ifrim DC, Saeed S, Jacobs C, van Loenhout J, de Jong D, Stunnenberg HG, Xavier RJ, van der Meer JW, van Crevel R, Netea MG. Bacille Calmette-Guerin induces NOD2-dependent nonspecific protection from reinfection via epigenetic reprogramming of monocytes. Proc Natl Acad Sci U S A. 2012 Oct 23;109(43):17537-42. doi: 10.1073/pnas.1202870109. Epub 2012 Sep 17. PMID 22988082
- [Background] Brandau S, Riemensberger J, Jacobsen M, Kemp D, Zhao W, Zhao X, Jocham D, Ratliff TL, Bohle A. NK cells are essential for effective BCG immunotherapy. Int J Cancer. 2001 Jun 1;92(5):697-702. doi: 10.1002/1097-0215(20010601)92:53.0.co;2-z. PMID 11340575
- [Background] Rusek P, Wala M, Druszczynska M, Fol M. Infectious Agents as Stimuli of Trained Innate Immunity. Int J Mol Sci. 2018 Feb 3;19(2):456. doi: 10.3390/ijms19020456. PMID 29401667
- [Background] Bekkering S, Blok BA, Joosten LA, Riksen NP, van Crevel R, Netea MG. In Vitro Experimental Model of Trained Innate Immunity in Human Primary Monocytes. Clin Vaccine Immunol. 2016 Dec 5;23(12):926-933. doi: 10.1128/CVI.00349-16. Print 2016 Dec. PMID 27733422
- [Background] Yamazaki-Nakashimada MA, Unzueta A, Berenise Gamez-Gonzalez L, Gonzalez-Saldana N, Sorensen RU. BCG: a vaccine with multiple faces. Hum Vaccin Immunother. 2020 Aug 2;16(8):1841-1850. doi: 10.1080/21645515.2019.1706930. Epub 2020 Jan 29. PMID 31995448
- See also: official report of the coronavirus in colombia — http://www.ins.gov.co/Noticias/Paginas/Coronavirus.aspx